CLINICAL TRIAL: NCT01045525
Title: Prospective Randomized Study Comparing the Effect of Phlebotomy and Lifestyle and Diet Advices vs Lifestyle and Diet Advices Only on Glycemia in Patients With Dysmetabolic Liversiderosis
Brief Title: Phlebotomy and Lifestyle and Diet Advices vs Lifestyle and Diet Advices Only in Patients With Dysmetabolic Liversiderosis
Acronym: SAIGNEES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUDRACT 2009-A00831-56; PHRC / 09-02 (Other: Sponsor)
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Liver Cirrhosis; Iron Overload
Keywords: Phlebotomy; Dysmetabolic liversiderosis; Hepatic Iron overload
MeSH Terms: conditions — Liver Cirrhosis; Iron Overload | interventions — Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phlebotomy + lifestyle and diet advices (Experimental)
  Interventions: Procedure: Phlebotomy
- Lifestyle and diet advices (Active Comparator)
  Interventions: Behavioral: Lifestyle and diet advices

INTERVENTIONS:
Procedure: Phlebotomy — From 300 to 400mL for women; From 350 to 450mL for men
  Other Names: Non applicable
  Arms: Phlebotomy + lifestyle and diet advices
Behavioral: Lifestyle and diet advices — 2 Booklets with Dietary and physical activity advices
  Other Names: Non applicable
  Arms: Lifestyle and diet advices

SUMMARY:
Insulin resistance-associated hepatic iron overload (IR-HIO), also defined as dysmetabolic iron overload syndrome or dysmetabolic liversiderosis, is a common cause or iron overload in France, mainly in middle-age patients with increased serum ferritin levels associated with normal serum transferrin saturation, and normal serum iron concentration in the absence of other known cause of increased serum ferritin levels.

Treatment includes a combination of dietary measures and physical activity to correct metabolic disorders. Phlebotomies seem to be beneficial when serum ferritin level is high.

This study aims at comparing the effect of iron depletion (by phlebotomy) plus lifestyle and diet advices versus lifestyle and diet advices alone on blood glucose level and insulin sensitivity in subjects with IR-HIO in order to assess the benefits of phlebotomies on the reduction of risk of diabetes and cardiovascular associated complications.

DETAILED DESCRIPTION:
Non applicable

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Signed written informed consent
* Ferritin ≥ 450 µg/L and ≤ 1500 µg/L
* Hepatic iron overload proved by MRI or histological biochemical measurement (Iron hepatic concentration ≥ 50 μmol/g)
* At least one of the following criteria :

  * Body mass index > 25 kg/m²
  * Systolic blood pressure ≥ 140mmHg or diastolic blood pressure ≥ 90 mmHg or antihypertensive treatment
  * Abdominal obesity (waist measurement ≥ 94 cm for men and ≥ 80 cm for women)
  * Fasting triglyceridemia ≥ 1.7 mmol/L or triglyceride-lowering treatment
  * Fasting HDL cholesterol < 1.03 mmol/L for men and < 1.29 mmol/L for women or HDL cholesterol-elevating treatment
  * Fasting blood glycemia ≥ 5.6 mmol/L

Exclusion Criteria:

* Subjects deprived of their liberty by judicial or administrative decision
* Pregnant women
* Other causes of increased serum ferritin levels:

  * Inflammatory syndrome (CRP >10 mg/L) or inflammatory, immune or malignant diseases
  * Hyper-hemolysis
  * Alcohol consumption more than 210 g for men and 140 g for women per week within the year before inclusion
  * Haemochromatosis established by the C282Y homozygous genotype
  * Chronic hepatic cytolysis due to : viral infection (HBV, HCV), alcohol, hyperthyroid disease, celiac disease, drug or immune hepatitis
  * Increased serum ferritin levels - cataract syndrome (familial cataract or personal history of cataract before 50 years of age)
  * Low ceruloplasmin level
  * Porphyria (cutaneous signs)
* Contraindication of phlebotomy

  * Haemoglobin <13 g/dL for men and <12g/dL for women (threshold established by the French Blood Agency)
  * Congestive heart failure or coronary heart disease
  * Hepatic failure (TP<60%), renal failure (GFR <50mL/min) or respiratory insufficiency (chronic dyspnea)
  * Poor venous system
* Fasting blood glycemia > 7 mmol/L or type 1 or type 2 diabetes, treated or not
* Use of drugs known to have anti-steatotic effects : metformin, thiazolidinedione

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2010-01; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Fasting blood glycemia (T0 of Oral Glucose Tolerance Test) | 12 months

SECONDARY OUTCOMES:
Rate of Body mass index > 25 kg/m² | 12 months
Rate of systolic blood pressure ≥ 130mmHg or diastolic blood pressure ≥ 85 mmHg or antihypertensive treatment | 12 months
Rate of abdominal obesity (waist measurement ≥ 94 cm for men and ≥ 80 cm for women) | 12 months
Rate of fasting triglyceridemia ≥ 1.7 mmol/L or triglyceride-lowering treatment | 12 months
Rate of fasting HDL cholesterol < 1.03 mmol/L for men and < 1.29 mmol/L for women or HDL cholesterol-elevating treatment | 12 months
Rate of fasting glycemia ≥ 5.6 mmol/L | 12 months
HbA1c value | 12 months
Quality of life estimated with SF36 form and tolerance to treatment | 12 months
Insulinoresistance indexes calculated at T0 and T30 min of Oral Glucose Tolerance Test (OGTT) | 12 months
Biological markers: CRP, hyaluronic acid, fibrometer | 12 months
myocardial deformation | 12 months
  Two dimensional (2D) speckle tracking echocardiography (STE)

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice LAINE, MD, Principal Investigator — Rennes University Hospital; Eric BELLISSANT, MD, PhD, Study Chair — Rennes University Hospital
Locations (5):
- France (5):
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - La Roche Sur Yon Hospital, La Roche-sur-Yon
  - Lorient Hospital, Lorient
  - Service des maladies du foie - Hôpital Pontchaillou, Rennes
  - Saint-Malo Hospital, St-Malo

REFERENCES:
- [Result] Laine F, Ruivard M, Loustaud-Ratti V, Bonnet F, Cales P, Bardou-Jacquet E, Sacher-Huvelin S, Causse X, Beusnel C, Renault A, Bellissant E, Deugnier Y; Study Group. Metabolic and hepatic effects of bloodletting in dysmetabolic iron overload syndrome: A randomized controlled study in 274 patients. Hepatology. 2017 Feb;65(2):465-474. doi: 10.1002/hep.28856. Epub 2016 Nov 10. PMID 27685251